CLINICAL TRIAL: NCT03205930
Title: A Phase I/Ⅱ Open, Single Center, One-armed Trail, Neo - MASCT Treatment for Advanced NSCLC of the Safety and Efficacy.
Brief Title: Neo-MASCT Immunotherapy for Advanced NSCLC.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Collaborators: Hengrui Yuanzheng Bio-Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo-MASCT
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single center single arm clinical study
Masking Description: Open clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neo-MASCT (Experimental): Neoantigen Multiple Target Antigen Stimulating Cell Therapy ( Neo-MASCT)
  Interventions: Biological: Neo-MASCT

INTERVENTIONS:
Biological: Neo-MASCT — The end product of Neo - MASCT technology is DC and CTL cells.DC injection,in each treatment cycle day 8, axillary, inguinal lymph node with subcutaneous injection. CTL cells， in every treatment cycle 21-28 days.

SUMMARY:
Neoantigen （Neo）is a new targets for immune cells，that the DC neoantigen immunotherapy was more effective in triggering specific T-cell responses. Neo-MASCT using the DC vaccine and neoantigen T cells .Dendritic cells(DC) was induced from autologous peripheral blood，and be loaded with antigens and re-infused. In vitro, antigen-pulsed DC can stimulate autologous T-cell proliferation and induction of autologous specific cytotoxic T-cells(CTL)，similarly re-infused.

The study is aimed to evaluate the safety of Neo-MASCT in patients with advanced NSCLC.

DETAILED DESCRIPTION:
This study is divided into two stages. The first stage is the safety study in small samples, and the second stage is the sample size expansion phase.

20 failed standard treatment patients with advanced or recurrent NSCLC will be recruited .

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18 to 80 years old.
2. The failure standard treatment subjects with advanced or relapsed NSCLC.
3. Informed consent of the patient/legal representative was signed.
4. Other anti-cancer treatments are at least one month apart from the study .
5. The eastern cancer cooperative group (ECOG) was rated 0-2.
6. According to the The reaction of solid tumors v1.1 (RECIST1.1 standard), there must be at least one measurable lesion .
7. The baseline blood and biochemical targets met the following criteria: The hemoglobin ≧ 85g/L ;White blood cells ≧ 3.0 x10 ^ 9 / L;Platelet ≧ 50 x10 ^ 9 / L;alanine aminotransferase (ALT), serum aspartate transaminase(AST) ≦ 2.5 times normal value limit; For patients with live metastases, ALT and AST are five times the normal limit; The alkaline phosphatase(ALP) ≦ 2.5 times the normal value; Serum bilirubin less than 1.5 times the normal value limit;

Exclusion Criteria:

1. Participate in the planning or implementation of the research .
2. In addition to other clinical studies, unless it is an observational clinical study .
3. Being pregnant or planning a pregnancy.
4. Refuse to provide a blood specimen .
5. Allergic to sodium hydroquinone .
6. There is a history of organ transplantation
7. Brain transfer of the active period
8. Immunosuppressant drugs are currently in use or within 14 days prior to treatment.
9. The following exceptions are:Nasal, inhaled, topical use of steroid, or topical steroids (such as interjoint injection) .
10. Use a corticosteroid, no more than 10mg/day of prednisolone or its equivalent .
11. The use of steroids as a preventative treatment for hypersensitivity (such as CT scans) .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 1 to 2 years
  The incidence of treatment-related adverse events were graded with the use of the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03

SECONDARY OUTCOMES:
Clinical response of treatment according to RESIST v1.1 criteria | 1 to 2 years
  Objective Response Rate (ORR)
Disease Control Rate (DCR) based on RESIST v1.1 criteria. | 1 to 2 years
  Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD).
Progression-Free Survival (PFS) based on RESIST v1.1 criteria. | From enrollment to progression of disease. Estimated about 6 months
  The length of time from enrollment until the time of progression of disease
Overall Survival (OS) based on RESIST v1.1 criteria. | From enrollment to death of patients
  The length of time from enrollment until the time to death
Elispot report | 1 to 2 years
  The relationship between clinical efficacy and antigen specific immune response

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaodong Jiang, Jiangsu, Doctor, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qiao Y, Hui K, Hu C, Wang M, Sun W, Liu L, Dong C, Jiang X. Efficacy and safety of PD-1 blockade-activated neoantigen specific cellular therapy for advanced relapsed non-small cell lung cancer. Cancer Immunol Immunother. 2025 Jan 3;74(2):60. doi: 10.1007/s00262-024-03906-z. PMID 39751937